CLINICAL TRIAL: NCT04314752
Title: Development of a Research Infrastructure for Understanding and Addressing Multiple Myeloma Disparities
Acronym: MEDULLA
Status: Recruiting | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Cancer Registry of Greater California (Unknown)
Responsible Party: Sponsor
Other Study IDs: 1487154
Record Dates: First submitted 2020-03-09; First posted 2020-03-19 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Study team will collect 2ml of saliva from participants who consent to the biospecimen collection portion of the study. Saliva will be used for genetic and genomic research
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of the proposed study are to develop and evaluate protocols for ethnic/racial minority-specific research using cancer registry data. In conjunction with the Cancer Registry of Greater California (CRGC), the investigators have developed procedures to identify, recruit, and survey ethnic/racial minority patients with MM. To pilot the study, the investigators aim initially to test the feasibility of this protocol by contacting 400 eligible patients (100 African Americans, 100 Latinos, 100 Asian American/Native Hawaiian/Pacific Islander-AANHPI and 100 non-Hispanic Whites as a comparison group) to conduct a pilot survey through which will ascertain etiological and survival-related factors for MM. Ultimately, the investigators hope the findings from this pilot will yield insight into the best practices for recruiting minorities with MM and serve as the basis for larger population-based studies of MM etiology and survival.

The next phase of this study is to expand the study to all 3 California Cancer Registries, including the Greater Bay Area Cancer Registry and the Los Angeles Cancer Surveillance Program and Cancer Registry of Greater California. We will increase the sample size to recruit atleast 1000 participants per racial/ethnic group. We will also request to increase the scope of the study to also continue a survivorship cohort.

DETAILED DESCRIPTION:
Eligible patients will include AAs, Latinos and AANHPIs who were diagnosed with a first primary, pathologically confirmed MM within the previous five years and who were at least 21 years of age at the time of diagnosis. We will also include, as a comparison group, non-Hispanic White patients. Patients must have been diagnosed in one of counties of California. Patients must be alive at the time of study and able to provide informed consent. We will not include those who are unable to consent, pregnant women, or prisoners.

Initially, in the pilot phase, we randomly selected 100 eligible patients from each race/ethnicity mentioned above to participate in the pilot study. As the pilot has been completed, we now aim to contact at recruit 1,000 patients per race/ethnic group reported to all three population cancer registries in the state, including the Greater Bay Area Cancer Registry and the Los Angeles Cancer Surveillance Program and Cancer Registry of Greater California until 2025. Patients diagnosis dates for the next phase of the study (June 2021-May 2025) will include diagnosis dates from 2018-2023, as there is a 2 year lag between patients cancer diagnosis and cancer registries information recorded.

Drs. Carvajal-Carmona and Cress have coordinated with MEDULLA investigators and CRGC research staff to develop a questionnaire for racial/ethnic minorities with Multiple Myeloma. The survey focuses on demographics, risk factors, cancer treatment, quality of life, and social determinants of health. All survey items are adapted from previously tested and validated surveys. The survey is expected to take approximately 30-45 minutes to complete.

CRGC staff, under Dr. Cress supervision, will identify eligible participants using the criteria described above based on diagnostic information in the CRGC database. The research team will be following California Cancer Registry policies and procedures for release of data. CRGC staff will extract patients contact information from the registry and will provide this information to research staff at UC Davis, who will work under Dr. Carvajal-Carmona's supervision.

The UC Davis Research team will initially mail each eligible participants a postcard and a survey study packet that will include: 1) Simple instruction sheet 2) An introductory letter that details the study 3) Information sheet that details on informed consent 4) Survey instruction sheet 5) A paper copy of the survey 5) Incentive selection sheet and option to continue to the second part of study 6) Brochures about the cancer registry and the UC Davis Comprehensive Cancer Center, and return pre-paid envelope.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a first primary pathologically confirmed case of Multiple Myeloma within the previous 5 years
* At least 21 years of age at the time of diagnosis
* Must have been diagnosed in one of the 48 counties in California
* Participant must be alive
* Identify as one of the following: African American, Latino, Asian American/Native Hawaiian/Pacific Islander, Non-Hispanic White

Exclusion Criteria:

* People who have not been diagnosed with Multiple Myeloma
* Under the age of 21
* Pregnant
* Prisoner

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will recruit 4,000 participants (1000 Latinos/ 1000 African Americans/ 1000 Asian American/Native Hawaiian/Pacific Islanders/ 1000 Non-Hispanic Whites). Participants will be randomly selected from cancer registry using the criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Review the response rate of mailed out surveys, compared by race/ethnicity and disease status | 2025
  Response Rate in percentage
Response rate for saliva kits compared to survey response and determine if there is a disparity in participation between race/ethnic groups | 2025
  Response Rates in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Luis Carvajal-Carmona, PhD, Principal Investigator — University of California, Davis; Rosemary Cress, DrPh MPH, Principal Investigator — Cancer Registry of California
Locations (1):
- University of California Davis Comprehensive Cancer Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No
Once everything is de-identified, we may share data or genetic information with dbGaP, a database of genotypes and phenotypes through the NIH for additional research. Protocols for additional research will be submitted to IRB for approval before use of this data or genetic information.

DOCUMENTS (2):
  • Study Protocol (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT04314752/Prot_000.pdf
  • Informed Consent Form (2019-12-02): https://cdn.clinicaltrials.gov/large-docs/52/NCT04314752/ICF_001.pdf